CLINICAL TRIAL: NCT04931823
Title: A Phase 1, Multicenter, Single Agent Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of CPO-100 in Adult Patients With Advanced Solid Tumors
Brief Title: Dose Escalation and Dose Expansion Study of CPO-100 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Conjupro Biotherapeutics, Inc. (Industry)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPO-100-US-101
Record Dates: First submitted 2021-06-04; First posted 2021-06-18 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor
Keywords: Breast Cancer; Prostate Cancer; Gastric Cancer; Lung Cancer; Head and Neck Cancer; Ovarian Cancer; Docetaxel; Docetaxel albumin-bound; DTX-HSA; CPO-100; Phase 1; Taxane Naïve; Solid Tumor; Stage 4; Metastatic Cancer; Cancer; Advanced Cancer; Taxane; Non-resectable tumor
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Stomach Neoplasms; Lung Neoplasms; Head and Neck Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Intervention Model Description: Modified "3+3" dose escalation design followed by dose expansion at the MTD (maximum tolerated dose).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A-1: Dose Escalation (Experimental): CPO-100 administered intravenously in cycles of 3 weekly doses with 1 week rest (1 cycle = 4 weeks).
  Interventions: Drug: CPO-100
- Part A-2: Dose escalation (Experimental): CPO-100 administered intravenously in cycles of 3 weekly doses with 1 week rest (1 cycle = 4 weeks) with the option to administer G-CSF in cycle one. Starting dose will be 45 mg/m2.
  Interventions: Drug: CPO-100
- Part B: Cohort 1 (Experimental): CPO-100 administered intravenously in cycles of 3 weekly doses with 1 week rest (1 cycle = 4 weeks) at the recommended Phase 2 dose (X mg/m2) in 15 patients with taxane naïve advanced solid tumors of gastric, head and neck, lung, and ovarian.
  Interventions: Drug: CPO-100
- Part B: Cohort 2 (Experimental): CPO-100 administered intravenously in cycles of 3 weekly doses with 1 week rest (1 cycle = 4 weeks) at the recommended Phase 2 dose (X mg/m2) in 15 patients with taxane naïve advanced breast cancer.
  Interventions: Drug: CPO-100
- Part B: Cohort 3 (Experimental): CPO-100 administered intravenously in cycles of 3 weekly doses with 1 week rest (1 cycle = 4 weeks) at the recommended Phase 2 dose (X mg/m2) in 15 patients with taxane naïve advanced prostate cancer.
  Interventions: Drug: CPO-100
- Part B: Cohort 4 (Experimental): CPO-100 administered intravenously in cycles of 3 weekly doses with 1 week rest (1 cycle = 4 weeks) at the recommended Phase 2 dose (X mg/m2) in 15 patients with either ovarian or/and breast cancer who have failed prior taxane treatment (ie, either progressed on a taxane regimen or within 6 months of receiving a taxane regimen).
  Interventions: Drug: CPO-100

INTERVENTIONS:
Drug: CPO-100 — Docetaxel albumin-bound
  Other Names: DTX-HSA

SUMMARY:
This is a Phase 1, multicenter, open-label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, and preliminary evidence of antitumor activity of CPO-100 administered intravenously in cycles of 3 weekly doses with 1 week rest (1 cycle = 4 weeks) in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study has three parts. Part A-1 is a dose-escalation phase with a modified "3+3" design in patients with metastatic or unresectable advanced solid tumors to evaluate the safety, tolerability and pharmacokinetics (PK) as a single agent. Two patients will be enrolled at each of the first 2 dose levels and observed for safety during the first cycle. If there are no ≥Grade 2 treatment emergent adverse events (TEAE) that are clinically significant and attributed to the study drug as assessed by the investigator during Cycle 1 for any of the patients in the first two dose levels, the 3rd dose level and beyond will follow the traditional 3+3 design. Dose escalation during the "3+3" period for each subsequent cohort of patients will be guided by the incidence of CPO-100-related adverse events (AE) as graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) CTCAE v5.0 in the first 4 weeks of dosing [the Dose Limiting Toxicity (DLT) evaluation period].

In Part A-2, the starting dose for this part will be 45 mg/m2. This dose was established in Part A-1 as being that dose at which the use of Granulocyte-colony stimulating factor ()G-CSF is indicated given that the only Grade 3 treatment-related adverse events noted were related to neutropenia and was well managed with G-CSF support. Prophylactic use of G-CSF will be permitted in Cycle 1 based on the investigator judgement.

This additional intervention of primary prophylaxis will be explored in order to determine if the risk of febrile neutropenia (FN) under these circumstances is reduced. Dose escalation during the 3+3 period for each subsequent cohort of patients will be guided by the incidence of CPO-100-related adverse events (AE) as graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 in the first 4 weeks of dosing (the DLT evaluation period).

After the Maximum Tolerated Dose (MTD) of weekly dosing schedule has been established, a recommended Phase 2 dose will be selected based on evaluation of the PK, and safety and tolerability profile on all available Part A study data by the Safety Review Committee (SRC). The selection of the Recommended Phase 2 Dose (RP2D) will consider all available clinical and non-clinical CPO-100 data as well as relevant docetaxel published data.

Part B expansion phase will further evaluate the safety and tolerability as well as the preliminary antitumor activity at the selected RP2D. Four cohorts of patients are included in Part B:

* Cohort 1: taxane naïve advanced/metastatic gastric, head and neck, lung, and ovarian cancers
* Cohort 2: taxane naïve advanced/metastatic breast cancer
* Cohort 3: taxane naïve advanced /metastatic prostate cancer
* Cohort 4: advanced/metastatic breast or ovarian cancer who have either progressed on a taxane or have developed progressive disease within 6 months of receiving a taxane.

The taxane naïve patient population is defined as patients who have not received taxane or taxane-based therapies for their metastatic diseases or patients who had suboptimal taxane exposure defined as having received less than 2 cycles of taxane or taxane-based therapies due to intolerability for their metastatic diseases. Patients who have received taxane or taxane-based therapies for their neoadjuvant treatment or patients who have received taxane or taxane-based therapies for their adjuvant treatment without disease progression during treatment are also considered taxane naïve, as long as they have not received taxane or taxane-based therapies to treat the metastatic diseases.

It is estimated that approximately 60 patients can be enrolled in Parts A-1 and A-2. The exact number of patients will depend on the number of dose levels tested. A total of 60 patients, 15 patients in each cohort will be enrolled in Part B.

The total duration of the study is estimated to be approximately 5 years. Patients may continue receiving CPO-100 until criteria for withdrawal are met. Patients deriving clinical benefit may continue to receive study medication for as long as they are benefiting from treatment. In the event the study closes or terminates while patients are still benefiting from and receiving CPO-100, every effort will be made to continue drug supply.

ELIGIBILITY:
Inclusion Criteria - Parts A-1, A-2, and B:

1. Presence of a pathologically documented (histology or cytology) locally advanced or metastatic solid tumor cancer.
2. Patients has failed at least 2 lines of conventional systemic therapy or have no other standard of care therapies available for their cancer. Prostate cancer patients should have received adenosine triphosphate (ADT) alone,(GnRH agonist, GnRH antagonist, or surgical orchiectomy and a pathway targeted agent such as abiraterone, enzalutamide, etc (castration-resistant prostate cancer). M1 disease must be present (not just biochemical recurrence).
3. Male or female patients18 years of age or older.
4. ECOG (Eastern Cooperative Oncology Group) performance status (PS) of 0, 1 or 2
5. Having at least one measurable target lesion present and documented by RECIST 1.1 for each cancer other than prostate cancer. Patients with prostate cancer may be enrolled with non-measurable disease providing the patient with a prostate-specific antigen (PSA) increase that is ≥25% and ≥2 ng/mL above the nadir, which is confirmed by a second value ≥3 weeks later, or 2 or more new bone lesions on imaging.
6. Adequate major system function defined as:

   1. Bone marrow reserve:

      Absolute neutrophil count (ANC) ≥1.5 x109/L Platelet count ≥ 100 x109/L Hemoglobin ≥9 g/dL without transfusion (the patient needs to be transfusion independent)
   2. Hepatic function:

      Total bilirubin ≤ upper limit of normal (ULN) (unless the subject has Grade 1 bilirubin elevation due to Gilbert's disease or a similar syndrome involving slow conjugation of total bilirubin); And aspartate aminotransferase (AST) / serum glutamic oxaloacetic transaminase (SGOT) and/or alanine aminotransferase (ALT) / serum glutamic pyruvic transaminase (SGPT) ≤ 1.5 x ULN with alkaline phosphatase ≤2.5 x ULN.
   3. Renal function:

      Normal serum creatinine ≤1.5 mg/dL (133 μmol/L) OR calculated creatinine clearance ≥50 mL/min. (Cockcroft - Gault formula)
   4. Coagulation:

   Adequate coagulation parameters defined as International Normalization Ratio (INR) ≤2.
7. Adequate methods of contraception for female patients of reproductive potential during the study and for at least 6 months following last dose. Male patients with female partners of childbearing potential and women patients of childbearing potential are required to use two forms of acceptable contraception, including 1 barrier method, during their participation in the study and for at least 3 months following last dose. Male patients must also refrain from donating sperm during their participation in the study.
8. Life expectancy ≥3 months.
9. Willingness and ability to comply with study and follow-up procedures.
10. Ability to understand the nature of this study and give written informed consent.

Additional Inclusion Criteria for the dose expansion cohort - Part B

1. Pathologically confirmed (histology or cytology) of the following cancer types:

   1. Cohort 1: taxane naïve advanced/metastatic gastric cancer, lung cancer, head and neck cancer, or ovarian cancer;
   2. Cohort 2: taxane naïve advanced/metastatic breast cancer;
   3. Cohort 3: taxane naïve advanced/metastatic prostate cancer.
   4. Cohort 4: advanced/metastatic breast or ovarian cancer patients who have either progressed on a taxane or have developed progressive disease within 6 months of receiving a taxane;
2. With the exception of Cohort 4 above, taxane naïve patients must not have received taxane or taxane based therapies for their metastatic diseases. Patients who had suboptimal taxane exposure defined as having received less than 2 cycles of taxane or taxane based therapies due to intolerability for their metastatic diseases, patients who have received taxane or taxane based therapies for their neoadjuvant treatment or patients who have received taxane or taxane based therapies for their adjuvant treatment without disease progression during treatment are also considered taxane naïve, as long as they have not received taxane or taxane based therapies to treat the metastatic diseases.

Exclusion Criteria - Part A and B

1. Most recent chemotherapy ≤14 days or have residual NCI CTCAE greater than Grade 1 chemotherapy-related side effects, with the exception of alopecia.
2. Use of any experimental drug ≤28 days or 5 half-lives (whichever is shorter) prior to the first dose of CPO-100. For study drugs for which 5 half-lives is ≤28 days, a minimum of 14 days between termination of the study drug and administration of CPO-100 is required.
3. Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89 and lutetium 177) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
4. Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
5. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 2 weeks previously and there is no evidence of central nervous system disease progression, and no requirement for chronic corticosteroid therapy.
6. Leptomeningeal metastases or spinal cord compression due to disease.
7. Known serious hypersensitivity reactions to docetaxel or life-threatening toxicity due to prior exposure to docetaxel
8. Pregnant or lactating.
9. Acute or chronic liver, renal, or pancreatic disease that in the opinion of the investigator would put the patient at unjustified increased risk by participating in this study or could interfere with the interpretation of the study results.
10. Other systemic disease that in the opinion of the investigator would put the patient at unjustified increased risk by participating in this study or could interfere with the interpretation of the study results.
11. Any of the following cardiac diseases currently or within the last 6 months:

    * Left ventricular ejection fraction (LVEF) <50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
    * Corrected QT (QTc) interval >470 ms (average of 3 tracings) on screening electrocardiogram (ECG)
    * Unstable angina pectoris
    * Congestive heart failure according to the New York Heart Association (NYHA) ≥ Grade 2)
    * Acute myocardial infarction
    * Conduction abnormality not controlled with pacemaker or medication
    * Significant ventricular or supraventricular arrhythmias. (Patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible.)
12. Inadequately controlled hypertension (ie, systolic blood pressure (SBP) >180 mmHg or diastolic blood pressure (DBP) >100 mmHg). Subjects with values above these levels must have their blood pressure (BP) controlled with medication prior to starting treatment.
13. Serious active infection at the time of treatment, or another serious underlying medical condition that that in the judgment of the investigator would impair the ability of the patient to receive protocol treatment.
14. HIV positive test within 8 weeks of screening. HIV positive patients with T-cell (CD4+) counts ≥350 cells/mL and not receiving treatment or does not plan to be treated with antiretroviral medication will be eligible for the study. Testing for seropositive status during screening will be at the discretion of the investigator in patients without previously reported results.
15. Active hepatitis B, or hepatitis C infection.

    * Patients will be tested for hepatitis C virus (HCV) and hepatitis B virus (HBV) at Screening.
    * Patients with hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA level is below the limit of detection by PCR) may be enrolled into the study. Subjects with controlled infections must undergo periodic monitoring of HBV DNA per treating physician.
    * Patients with hepatitis C (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) may be enrolled into the study. Patients with controlled infections must undergo periodic monitoring of HCV RNA per treating physician.
16. Presence of other active cancers, or history of treatment for invasive cancer ≤3 years. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (ie, non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
17. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
18. Routine use of corticosteroids or erythrocyte-stimulating factors as well as prophylactic use of colony-stimulating factors.
19. Use of any strong CYP3A4 inhibitor or strong inducer drugs ≤28 days or 5 half-lives (whichever is shorter) prior to the first dose of CPO-100. For CYP3A4 inducer drugs for which 5 half-lives is ≤28 days, a minimum of 14 days between discontinuation of the drug and administration of CPO-100 is required.
20. Use of herbal preparations/medications including, but are not limited to: St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. A minimum of 14 days between discontinuation of the herbal preparation/medications and administration of CPO-100 is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Part A-1: Number of subjects with Dose Limiting Toxicities (DLTs) | At the end of cycle 1 (each cycle is 28 days)
  Incidence of dose-limiting toxicities (DLT) during the DLT evaluation period. DLTs assessed per CTCAE v5.0, include grade ≥ 4 neutropenia, thrombocytopenia, anemia; grade ≥ 3 febrile neutropenia, nausea, vomiting, diarrhea, skin rash, fatigue, infusion reaction; any other grade ≥ 2 non-hematologic toxicity judged to be dose limiting; and treatment delay >14 days due to unresolved toxicities.
Part A-2: Number of subjects with Dose Limiting Toxicities (DLTs) when prophylactic use of G-CSF is allowed during Cycle 1 | At the end of cycle 1 (each cycle is 28 days)
  Incidence of dose-limiting toxicities (DLT) during the DLT evaluation period. DLTs assessed per CTCAE v5.0, include grade ≥ 4 neutropenia, thrombocytopenia, anemia; grade ≥ 3 febrile neutropenia, nausea, vomiting, diarrhea, skin rash, fatigue, infusion reaction; any other grade ≥ 2 non-hematologic toxicity judged to be dose limiting; and treatment delay >14 days due to unresolved toxicities.
Part B: Dose Expansion - Incidence and severity of Adverse Events | Screening to up to 4 years
  Incidence and severity of Adverse Events per CTCAE v5.0, including changes of Clinical Laboratory Values, Physical Exams, Vital Signs, Weight, Eastern Cooperative Oncology Group (ECOG) and ECG from baseline. Dosing delays and dosing intensity.

SECONDARY OUTCOMES:
Area Under the Curve (AUC0-t) for CPO-100 | 0, .5, 1, 2, 3, 4, 6, 8, 24, 48 and 72 hours (Day1) and Day 15
  Area under the plasma concentration curve (AUC0-t) will be from time zero to last quantifiable concentration.
Area Under the Curve (AUC0-∞) for CPO-100 | 0, .5, 1, 2, 3, 4, 6, 8, 24, 48 and 72 hours (Day1)
  Area under the plasma concentration curve (AUC0-∞) will be from time zero to infinity.
Cmax for CPO-100 | 0, .5, 1, 2, 3, 4 6, 8, 24, 48 and 72 hours (Day 1) and Day 15
  Cmax will be estimated from the maximum post-dose concentration recorded for each patient.
Tmax for CPO-100 | Time Frame: 0, .5, 1, 2, 3, 4 6, 8, 24, 48 and 72 hours (Day 1) and Day 15
  Tmax will be estimated from the relative time of the maximum post-dose concentration recorded for each patient.
Overall response rate (ORR) | At the end of every 28 day cycle for up to 4 years
  The proportion of patients achieving a partial response (PR) or complete response (CR) per RECIST 1.1 supplemented by recommendations from the Prostate Cancer Clinical Trials Working Group 3 (PCCTWG3).
Disease control rate (DCR) | At the end of every 28 day cycle for up to 4 years
  The proportion of patients achieving a stable disease (SD), PR, CR per RECIST 1.1 supplemented by recommendations from the Prostate Cancer Clinical Trials Working Group 3 (PCCTWG3).
Duration of Response (DoR) | From first PR or CR until disease progression or death up to 4 years
  Time from first PR or CR until progression of death using definition of PR and CR per (RECIST) 1.1 supplemented by recommendations from the Prostate Cancer Clinical Trials Working Group 3 (PCCTWG3).
Progression-Free Survival (PSF) | From first dose until documented disease progression or death up to 4 years
  Time from first dose until disease progression or death using RECIST 1.1 supplemented by recommendations from the Prostate Cancer Clinical Trials Working Group 3 (PCCTWG3) for progression.

CONTACTS AND LOCATIONS:
Overall Officials: Study Officials, Study Director — Conjupro Biotherapeutics, Inc.
Locations (8):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - The Cleveland Clinic Foundation, Lyndhurst, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Virginia Cancer Specialist, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Background] Aihara T, Kim Y, Takatsuka Y. Phase II study of weekly docetaxel in patients with metastatic breast cancer. Ann Oncol. 2002 Feb;13(2):286-92. doi: 10.1093/annonc/mdf027. PMID 11886007
- [Background] Andre N, Carre M, Pasquier E. Metronomics: towards personalized chemotherapy? Nat Rev Clin Oncol. 2014 Jul;11(7):413-31. doi: 10.1038/nrclinonc.2014.89. Epub 2014 Jun 10. PMID 24913374
- [Background] Aston WJ, Hope DE, Cook AM, Boon L, Dick I, Nowak AK, Lake RA, Lesterhuis WJ. Dexamethasone differentially depletes tumour and peripheral blood lymphocytes and can impact the efficacy of chemotherapy/checkpoint blockade combination treatment. Oncoimmunology. 2019 Jul 13;8(11):e1641390. doi: 10.1080/2162402X.2019.1641390. eCollection 2019. PMID 31646089
- [Background] Bruno R, Olivares R, Berille J, Chaikin P, Vivier N, Hammershaimb L, Rhodes GR, Rigas JR. Alpha-1-acid glycoprotein as an independent predictor for treatment effects and a prognostic factor of survival in patients with non-small cell lung cancer treated with docetaxel. Clin Cancer Res. 2003 Mar;9(3):1077-82. PMID 12631610
- [Background] de Wit R, de Bono J, Sternberg CN, Fizazi K, Tombal B, Wulfing C, Kramer G, Eymard JC, Bamias A, Carles J, Iacovelli R, Melichar B, Sverrisdottir A, Theodore C, Feyerabend S, Helissey C, Ozatilgan A, Geffriaud-Ricouard C, Castellano D; CARD Investigators. Cabazitaxel versus Abiraterone or Enzalutamide in Metastatic Prostate Cancer. N Engl J Med. 2019 Dec 26;381(26):2506-2518. doi: 10.1056/NEJMoa1911206. Epub 2019 Sep 30. PMID 31566937
- [Background] Gradishar WJ. Taxanes for the treatment of metastatic breast cancer. Breast Cancer (Auckl). 2012;6:159-71. doi: 10.4137/BCBCR.S8205. Epub 2012 Oct 25. PMID 23133315
- [Background] Hardin C, Shum E, Singh AP, Perez-Soler R, Cheng H. Emerging treatment using tubulin inhibitors in advanced non-small cell lung cancer. Expert Opin Pharmacother. 2017 May;18(7):701-716. doi: 10.1080/14656566.2017.1316374. Epub 2017 Apr 17. PMID 28388240
- [Background] Harvey V, Mouridsen H, Semiglazov V, Jakobsen E, Voznyi E, Robinson BA, Groult V, Murawsky M, Cold S. Phase III trial comparing three doses of docetaxel for second-line treatment of advanced breast cancer. J Clin Oncol. 2006 Nov 1;24(31):4963-70. doi: 10.1200/JCO.2005.05.0294. Epub 2006 Oct 10. PMID 17033039
- [Background] Minami H, Kawada K, Sasaki Y, Igarashi T, Saeki T, Tahara M, Itoh K, Fujii H. Pharmacokinetics and pharmacodynamics of protein-unbound docetaxel in cancer patients. Cancer Sci. 2006 Mar;97(3):235-41. doi: 10.1111/j.1349-7006.2006.00166.x. PMID 16542221
- [Background] Ohbatake Y, Fushida S, Tsukada T, Kinoshita J, Oyama K, Hayashi H, Miyashita T, Tajima H, Takamura H, Ninomiya I, Yashiro M, Hirakawa K, Ohta T. Elevated alpha1-acid glycoprotein in gastric cancer patients inhibits the anticancer effects of paclitaxel, effects restored by co-administration of erythromycin. Clin Exp Med. 2016 Nov;16(4):585-592. doi: 10.1007/s10238-015-0387-9. Epub 2015 Sep 10. PMID 26359244
- [Background] Palmeri L, Vaglica M, Palmeri S. Weekly docetaxel in the treatment of metastatic breast cancer. Ther Clin Risk Manag. 2008 Oct;4(5):1047-59. doi: 10.2147/tcrm.s3397. PMID 19209285
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579
- [Background] Socinski MA, Manikhas GM, Stroyakovsky DL, Makhson AN, Cheporov SV, Orlov SV, Yablonsky PK, Bhar P, Iglesias J. A dose finding study of weekly and every-3-week nab-Paclitaxel followed by carboplatin as first-line therapy in patients with advanced non-small cell lung cancer. J Thorac Oncol. 2010 Jun;5(6):852-61. doi: 10.1097/jto.0b013e3181d5e39e. PMID 20521351
- [Background] Urien S, Barre J, Morin C, Paccaly A, Montay G, Tillement JP. Docetaxel serum protein binding with high affinity to alpha 1-acid glycoprotein. Invest New Drugs. 1996;14(2):147-51. doi: 10.1007/BF00210785. PMID 8913835
- [Background] American Cancer Society. https://www.cancer.org/cancer/pancreatic-cancer/about/key-statistics.html Accessed 17 May 2022
- [Background] Deeken JF, Slack R, Weiss GJ, Ramanathan RK, Pishvaian MJ, Hwang J, Lewandowski K, Subramaniam D, He AR, Cotarla I, Rahman A, Marshall JL. A phase I study of liposomal-encapsulated docetaxel (LE-DT) in patients with advanced solid tumor malignancies. Cancer Chemother Pharmacol. 2013 Mar;71(3):627-33. doi: 10.1007/s00280-012-2048-y. Epub 2012 Dec 30. PMID 23274395
- [Background] Eheman C, Henley SJ, Ballard-Barbash R, Jacobs EJ, Schymura MJ, Noone AM, Pan L, Anderson RN, Fulton JE, Kohler BA, Jemal A, Ward E, Plescia M, Ries LA, Edwards BK. Annual Report to the Nation on the status of cancer, 1975-2008, featuring cancers associated with excess weight and lack of sufficient physical activity. Cancer. 2012 May 1;118(9):2338-66. doi: 10.1002/cncr.27514. Epub 2012 Mar 28. PMID 22460733
- [Background] NCCN Guidelines Version 1.2022, Management of Neutropenia
- [Background] Pronk LC. Modulation of docetaxel treatment [dissertation], Rotterdam: Erasmus Universiteit; 1997
- [Background] Simard EP, Ward EM, Siegel R, Jemal A. Cancers with increasing incidence trends in the United States: 1999 through 2008. CA Cancer J Clin. 2012 Mar-Apr;62(2):118-28. doi: 10.3322/caac.20141. Epub 2012 Jan 4. PMID 22281605
- [Background] Smith BD, Smith GL, Hurria A, Hortobagyi GN, Buchholz TA. Future of cancer incidence in the United States: burdens upon an aging, changing nation. J Clin Oncol. 2009 Jun 10;27(17):2758-65. doi: 10.1200/JCO.2008.20.8983. Epub 2009 Apr 29. PMID 19403886
- [Background] StatBite. U.S. pancreatic cancer rates. J Natl Cancer Inst. 2010 Dec 15;102(24):1822. doi: 10.1093/jnci/djq517. Epub 2010 Dec 7. No abstract available. PMID 21139097
- [Background] Sweeney CJ, Chen YH, Carducci M, Liu G, Jarrard DF, Eisenberger M, Wong YN, Hahn N, Kohli M, Cooney MM, Dreicer R, Vogelzang NJ, Picus J, Shevrin D, Hussain M, Garcia JA, DiPaola RS. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer. N Engl J Med. 2015 Aug 20;373(8):737-46. doi: 10.1056/NEJMoa1503747. Epub 2015 Aug 5. PMID 26244877
- [Background] Taxotere® US Package Insert (version 11/2021)
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Worni M, Guller U, White RR, Castleberry AW, Pietrobon R, Cerny T, Gloor B, Koeberle D. Modest improvement in overall survival for patients with metastatic pancreatic cancer: a trend analysis using the surveillance, epidemiology, and end results registry from 1988 to 2008. Pancreas. 2013 Oct;42(7):1157-63. doi: 10.1097/MPA.0b013e318291fbc5. PMID 23867367
- See also: Phase II study of weekly docetaxel in patients with metastatic breast cancer — https://pubmed.ncbi.nlm.nih.gov/11886007/
- See also: Metronomics: towards personalized chemotherapy? — https://pubmed.ncbi.nlm.nih.gov/24913374/
- See also: Dexamethasone differentially depletes tumour and peripheral blood lymphocytes and can impact the efficacy of chemotherapy/checkpoint blockade combination treatment — https://pubmed.ncbi.nlm.nih.gov/31646089/
- See also: Alpha-1-acid glycoprotein as an independent predictor for treatment effects and a prognostic factor of survival in patients with non-small cell lung cancer treated with docetaxel — https://pubmed.ncbi.nlm.nih.gov/12631610/
- See also: Cabazitaxel versus Abiraterone or Enzalutamide in Metastatic Prostate Cancer — https://pubmed.ncbi.nlm.nih.gov/31566937/
- See also: Taxanes for the treatment of metastatic breast cancer — https://pubmed.ncbi.nlm.nih.gov/23133315/
- See also: Emerging treatment using tubulin inhibitors in advanced non-small cell lung cancer — https://pubmed.ncbi.nlm.nih.gov/28388240/
- See also: Phase III trial comparing three doses of docetaxel for second-line treatment of advanced breast cancer — https://pubmed.ncbi.nlm.nih.gov/17033039/
- See also: Pharmacokinetics and pharmacodynamics of protein-unbound docetaxel in cancer patients — https://pubmed.ncbi.nlm.nih.gov/16542221/
- See also: Elevated alpha1-acid glycoprotein in gastric cancer patients inhibits the anticancer effects of paclitaxel, effects restored by co-administration of erythromycin — https://pubmed.ncbi.nlm.nih.gov/26359244/
- See also: Weekly docetaxel in the treatment of metastatic breast cancer — https://pubmed.ncbi.nlm.nih.gov/19209285/
- See also: A dose finding study of weekly and every-3-week nab-Paclitaxel followed by carboplatin as first-line therapy in patients with advanced non-small cell lung cancer — https://pubmed.ncbi.nlm.nih.gov/20521351/
- See also: Docetaxel serum protein binding with high affinity to alpha 1-acid glycoprotein — https://pubmed.ncbi.nlm.nih.gov/8913835/
- See also: A phase I study of liposomal-encapsulated docetaxel (LE-DT) in patients with advanced solid tumor malignancies — http://pubmed.ncbi.nlm.nih.gov/23274395/
- See also: Annual Report to the Nation on the status of cancer, 1975-2008, featuring cancers associated with excess weight and lack of sufficient physical activity — https://pubmed.ncbi.nlm.nih.gov/22460733/
- See also: Cancers with increasing incidence trends in the United States: 1999 through 2008 — https://pubmed.ncbi.nlm.nih.gov/22281605/
- See also: Future of cancer incidence in the United States: burdens upon an aging, changing nation — https://pubmed.ncbi.nlm.nih.gov/19403886/
- See also: U.S. pancreatic cancer rates — https://pubmed.ncbi.nlm.nih.gov/21139097/
- See also: Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer — https://pubmed.ncbi.nlm.nih.gov/26244877/
- See also: Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial — https://pubmed.ncbi.nlm.nih.gov/21969517/
- See also: Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine — https://pubmed.ncbi.nlm.nih.gov/24131140/
- See also: Modest improvement in overall survival for patients with metastatic pancreatic cancer: a trend analysis using the surveillance, epidemiology, and end results registry from 1988 to 2008 — https://pubmed.ncbi.nlm.nih.gov/23867367/